CLINICAL TRIAL: NCT03047616
Title: A Pilot Study to Develop Predictive Biomarkers for the Response to Immunotherapy in Lung Cancer
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 27516
Record Dates: First submitted 2017-02-06; First posted 2017-02-09 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of blood and urine specimens from patients receiving immunotherapy as part of their standard of care for the treatment of NSCLC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood and Urine Collection

SUMMARY:
Several immune checkpoint inhibitors targeting the PD-1 pathway have been developed with clinical trials showing an approximately 20% durable response in unselected patients with advanced non-small cell lung cancer (NSCLC). At the moment, no clear biomarker exists to accurately predict anti-PD1/PDL1 tumor responsiveness. The goal of this study is to broadly discover and evaluate the utility of blood based biomarkers for use in measuring and predicting response to immunotherapy in patients with lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Metastatic NSCLC
* Scheduled to initiate an immune checkpoint inhibitor
* Age >= 18 years
* Able to provide informed consent

Exclusion Criteria:

* Other, unrelated, concomitant active, invasive malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with non-small cell lung cancer (NSCLC)
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
the correlation between markers identified in the blood and in the primary tumor. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Charu Aggarwal, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Aggarwal C, Thompson JC, Chien AL, Quinn KJ, Hwang WT, Black TA, Yee SS, Christensen TE, LaRiviere MJ, Silva BA, Banks KC, Nagy RJ, Helman E, Berman AT, Ciunci CA, Singh AP, Wasser JS, Bauml JM, Langer CJ, Cohen RB, Carpenter EL. Baseline Plasma Tumor Mutation Burden Predicts Response to Pembrolizumab-based Therapy in Patients with Metastatic Non-Small Cell Lung Cancer. Clin Cancer Res. 2020 May 15;26(10):2354-2361. doi: 10.1158/1078-0432.CCR-19-3663. Epub 2020 Feb 26. PMID 32102950

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT03047616/Prot_SAP_000.pdf